CLINICAL TRIAL: NCT04867187
Title: Clinical Study of Repetitive Transcranial Magnetic Stimulation (RTMS) Efficacy Coupled With Mirror Therapy for Neuropathic Pain Relief
Brief Title: rTMS Efficacy Coupled With Mirror Therapy
Acronym: STIRM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21CH035; 2021-A00720-41 (Other: ANSM)
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Neuropathic Pain
Keywords: transcranial magnetic stimulation; virtual reality; mirror therapy; brain networks; predictive model
MeSH Terms: conditions — Neuralgia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Group 1: patient with 4 sessions of active mirror therapy followed by an rTMS stimulation session of the primary motor cortex (M1), Group 2: patient with 4 sessions of sham mirror therapy followed by rTMS of the primary motor cortex (M1).
Who Masked: Participant, Investigator
Masking Description: The (motor) task performed by the patient during the sham control mirror therapy session is identical to that performed in active mirror therapy. The only difference is that in sham mirror therapy there is no optical illusion of movement of the affected hand.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rTMS active and active mirror-based therapy using virtual reality (Experimental): The patient will have an amount of 4 sessions (S3, S5, S7 and S9) for 1.5 months: 1 session every 2 weeks. The patient will receive rTMS active and active mirror-based therapy using virtual reality.
  Interventions: Other: Repetitive transcranial magnetic stimulation (rTMS); Other: Mirror therapy using virtual reality
- rTMS active and sham mirror-based therapy using virtual reality (Sham Comparator): The patient will have an amount of 4 sessions (S3, S5, S7 and S9) for 1.5 months: 1 session every 2 weeks. The patient will receive rTMS active and sham mirror-based therapy using virtual reality.
  Interventions: Other: Repetitive transcranial magnetic stimulation (rTMS); Other: Mirror therapy using sham mirror

INTERVENTIONS:
Other: Repetitive transcranial magnetic stimulation (rTMS) — 20 minutes of high frequency (20Hz) rTMS.
Other: Mirror therapy using virtual reality — active mirror-based therapy
  Arms: rTMS active and active mirror-based therapy using virtual reality
Other: Mirror therapy using sham mirror — 20 minutes of sham mirror-based therapy
  Arms: rTMS active and sham mirror-based therapy using virtual reality

SUMMARY:
Neuropathic pain is particularly difficult to treat with classic first-line drugs. Neuromodulation techniques using repetitive transcranial magnetic stimulation (rTMS) are useful alternative, but there is a need to improve their analgesic effect.Virtual reality mirror therapy has shown the capacity to alleviate pain and may be easily coupled with rTMS.The present project will investigate in individuals with neuropathic pain the effects of the rTMS coupled with virtual reality mirror therapy.

DETAILED DESCRIPTION:
This project introduces a new research question that incorporates virtual reality mirror therapy into an established treatment protocol of repetitive transcranial magnetic stimulation (rTMS) for neuropathic pain relief. Neuropathic pain is particularly difficult to treat with classic first-line drugs. Neuromodulation techniques using repetitive transcranial magnetic stimulation (rTMS) are useful alternative, but there is a need to improve their analgesic effect.

Virtual reality mirror therapy has shown the capacity to alleviate pain and may be easily coupled with rTMS. The efficacy of using both techniques in neuropathic pain treatment is unknown. The present project will investigate in individuals with neuropathic pain the effects of the rTMS coupled with virtual reality mirror therapy on: 1) daily pain intensity (i.e. analgesic efficacy); 2) other components of pain and the quality of life; 3) brain activity.

It will be the first to provide insight into the efficacy of using together both non-invasive technics of cortical neuromodulation to alleviate pain.

ELIGIBILITY:
Inclusion Criteria:

* Clinical symptoms typical of neuropathic pain
* Refractory to drug therapies
* Lasting for at least 6 months, with a moderate to severe pain intensity (≥4/10 on Visual Analog Scale, VAS) and a stable pain treatment since 1month at least
* Having right to health benefits

Exclusion Criteria:

* Ferromagnetic components and implanted microprocessors (i.e. cochlear implants)
* Drug-resistant or active epilepsy, pacemaker, pregnancy, ongoing depression or personality troubles, and ongoing opioid treatment.
* Any other contraindications to MRI scanner (e.g., claustrophobia, etc.).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-10-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Pain intensity measurement | Week 9
  Averages of the daily visual analogue scale scores (min no pain max pain imaginable) measured during the first week (Week 1) and that measured during the week following the last session (week 9)

SECONDARY OUTCOMES:
Quality of life after treatment | week 12
  EQ5D scale (min = 0 worst imaginable health condition and max = 100 best health condition imaginable) and Analgesic consumption of Appeal
Spontaneous brain activity | week 12
  Functional MRI at rest
neuropathic dimension | Week 3, 5, 7, 9,12
  overall score of the neuropathic pain symptoms inventory (NPSI) (min = 0 no neuropathic pain and max = 100 intensive neuropathic pain)
Adverse events | Week 3, 5, 7, 9,12
  Nature and number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Roland Peyron, MDPHD, Principal Investigator — CENTRE HOSPITALIER DE SAINT-ETIENNE
Locations (2):
- France (2):
  - Hôpital Neurologique Pierre Wertheimer, Bron
  - Centre Hospitalier Universitaire de Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No